CLINICAL TRIAL: NCT04876716
Title: Azole-echinocandin Combination Therapy for Invasive Aspergillosis A Randomized Pragmatic Superiority Trial
Brief Title: Azole-echinocandin Combination Therapy for Invasive Aspergillosis
Acronym: IA-DUET
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: futility
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Principal Investigator, Bart Rijnders, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL72950.078.20; 2020-000627-40 (EudraCT Number)
Record Dates: First submitted 2021-04-14; First posted 2021-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Invasive Aspergillosis
Keywords: invasive aspergillosis; azole; echinocandin; combination therapy
MeSH Terms: interventions — Azoles; Voriconazole; isavuconazole; posaconazole; Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azole monotherapy (Active Comparator): Azole monotherapy
  Voriconazole or isavuconazole or posaconazole will be dosed according to the SPC and according to the route of administration (IV or orally) that is preferred by the treating physician. However, the dose may be changed based on therapeutic drug monitoring levels according to the local standard of care.
  Interventions: Drug: Azole
- Azole + Anidulafungin (Experimental): Azole + Anidulafungin
  Voriconazole or isavuconazole or posaconazole will be dosed according to the SPC and according to the route of administration (IV or orally) that is preferred by the treating physician. However, the dose may be changed based on therapeutic drug monitoring levels according to the local standard of care.
  Anidulafungin (Ecalta) is available as an intravenous formulation only. It will be used at the licensed dose of a 200mg loading dose on day 1 and 100mg QD thereafter. No dose adjustment is needed in patients with renal or hepatic insufficiency of any grade.
  Interventions: Drug: Azole; Drug: Anidulafungin

INTERVENTIONS:
Drug: Azole — Dosing according to the SPC
  Other Names: Voriconazole; isavuconazole; posaconazole
Drug: Anidulafungin — 200mg loading dose on day 1 and 100mg QD thereafter
  Other Names: Ecalta
  Arms: Azole + Anidulafungin

SUMMARY:
The goals of this study are 3-fold:

First, the main study and the primary endpoint will evaluate if the overall mortality can be decreased with initial azole-echinocandin combination therapy compared with triazole monotherapy in patients with IA and documented voriconazole susceptibility.

Second, the study design described will also allow to study several other subpopulations; Indeed, the outcome of the following subgroups will be evaluated as well; a. Patients starting azole monotherapy but who switch to directed therapy when it has become clear that the infection is caused by an azole resistant A. fumigatus. b. patients in which eventually no resistance data become available in relation to the treatment they received.

Third, the study will evaluate what the outcome is of patients that turn out to be infected with a triazole resistant A. fumigatus who started with a triazole-echinocandin combination therapy.

DETAILED DESCRIPTION:
Background of the study:

Patients with underlying haematological malignancies or immunocompromised for various other reasons, are prone to fungal infections. Invasive aspergillosis (IA) is a common complication during remission inducing chemotherapy for acute leukemia or other hematological malignancies, as well as those who have undergone allogeneic hematopoietic stem cell transplantation (HSCT) or solid organ transplantation (SOT).

For more than 15 years voriconazole, a drug of the triazole class, has been the recommended treatment for this life-threatening infection after a pivotal randomized trial showed an improved survival with voriconazole compared with amphotericin B deoxycholate. However, also with voriconazole the overall 6-week mortality is still unacceptably high at 25-30%.

Therefore, a randomized controlled trial assed the efficacy of voriconazole with or without anidulafungin for the treatment of IA in haematology patients to prove that combination therapy can improve outcome.Among the 277 patients with IA in this study, the 6-week mortality with combination therapy was 30% lower (19.3%) than with monotherapy (27.5%), p=0.087. In a post-hoc analysis of the 222 patients with radiographic abnormalities and a positive galactomannan antigen test, a statistically significant difference in mortality was observed (p=0.037). Though, this study did not result in conclusive evidence in favor of combination therapy, it is a credible study which adds to the already existing in vitro and animal studies in support of echinocandin triazole combination therapy for IA and thus paves the way for a second larger and pragmatic clinical trial. Another important and new consideration about the management of IA is the upcoming of infections with triazole-resistant A. fumigatus. This is increasingly becoming a worldwide problem and leads to longer hospital stay, higher costs and is associated with a very high mortality.

It is very likely that the excessive use of antifungals of the triazole class in agriculture has formed the basis of this problem.

Since 2018 the Dutch Working Party on Antibiotic therapy (SWAB) guideline on the management of invasive fungal infections therefore recommends upfront combination therapy (azole plus echinocandins or liposomal-amfotericine B) until resistance can be excluded as one of the treatment options for IA. Given the evidence in favor of voriconazole-echinocandin combination therapy as well as the increasing incidence of voriconazoleresistant A. fumigatus in Belgium and the Netherlands, a large clinical study on the value of combination therapy is urgently needed.

Objective of the study:

Primary objective

1. Evaluate if the survival in patients with a triazole susceptible IA can be improved when the initial therapy consists of triazole and echinocandin combination therapy instead of triazole monotherapy.

Secondary objectives

1. Evaluate if a triazole/echinocandin combination therapy improves the overall quality of life and if it is a cost-effective intervention
2. Evaluate the outcome of patients in which a triazole-resistant A. fumigatus is detected in relation to the initial antifungal therapy patients had received (i.e. triazole monotherapy or combination therapy).
3. Evaluate the outcome of patients in which resistance testing is unsuccessful in function of the antifungal therapy they received.
4. Evaluate if the baseline serum galactomannan value and the serum galactomannan kinetics are predictive of overall 6-week survival.

Study design:

A non-blinded phase 3 randomized pragmatic clinical trial.

Study population:

Immunocompromised patients who fulfill the EORTC/MSG host factor and mycological criteria of invasive aspergillosis ICU patients with influenza who fulfill a definition of IA specific for this population

Intervention:

Treatment with a triazole (voriconazole or isavuconazole or posaconazole) + anidulafungin IV. The triazole is administered for at least 6 weeks while anidulafungin is given for at least 7 and a maximum of 28 days.

Comparator:

Treatment with a triazole (voriconazole or isavuconazole or posaconazole) for at least 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Have started or will start voriconazole or isavuconazole (or posaconazole if voriconazole or isavuconazole cannot be given as per treating physician's decision) as antifungal therapy on the baseline visit.
3. For all patients: presence of one of the EORTC/MSG host factors as defined in appendix 1 or being admitted to the ICU with influenza
4. For non-ICU patients or ICU patients without influenza: Meet the EORTC/MSG clinical criterium (appendix 1)
5. For non-ICU patients or ICU patients without influenza: Meet the mycological criterium (appendix 1) or fulfil inclusion criterium 7
6. For ICU patients with influenza we consider an isolated positive sputum culture for Aspergillus spp. insufficient as amycological criterium. Therefore, in these patients only one of the following mycological criteria are acceptable; Serum galactomannan ≥0.5, BAL galactomannan ≥1.0 or Aspergillus spp. cultured in BAL fluid.
7. Please note that patients with AML receiving chemotherapy or patients with ALL receiving or having received corticosteroid therapy within the last 4 weeks in the context of their pre-phase, induction, consolidation, intensification or interphase treatment as well as patients receiving systemic immunosuppressive therapy for GVHD can be included before the mycological criterium is fulfilled on condition that they fulfill the EORTC/MSG lung CT radiology criteria (halo sign, well-described nodule, cavity as described in appendix 1) at the time of inclusion and as long as the mycological test results are expected to become available within 96 and no later than 7 days after inclusion. If these test results turn out to be negative, the patient will be withdrawn from the study and further treatment is at physician's discretion.
8. Written informed consent by patient or legal representative.

Exclusion Criteria:

1. Known history of allergy, hypersensitivity or serious reaction to azole or echinocandin antifungals;
2. Patients with chronic invasive aspergillosis or a chronic non-invasive aspergillus infection (e.g. aspergilloma) defined as the clinical or radiological sign of infection being present for >28 days.
3. Receipt of itraconazole, voriconazole, posaconazole or isavuconazole as prophylaxis for at least 7 days in the 14 days preceding the date of the first radiological signs of the Aspergillus infection. Patients in which the most recent serum level of the triazole given as prophylaxis was subtherapeutic can be included (*).
4. Receipt of echinocandin prophylaxis for >96 hours in the preceding 7 days
5. Receipt of systemic antifungal treatment with an echinocandin or an azole for the current episode of invasive aspergillosis for a duration of > 96 hours.
6. For patients in the Netherlands only: Diagnostic testing to exclude azole resistance will not be possible (sputum cultures are negative and BAL sampling will not be performed)
7. ICU patients only: Patients with a sequential organ failure assessment (SOFA) score >11 at the time of screening for the study are excluded. If randomization is done >24 hours after screening the calculation should be repeated before the patient can be randomized (appendix 3)
8. ICU patients only: Patients in which weaning from the ventilator or ECMO system is deemed unlikely due to irreversible lung damage
9. Patients with any condition which, in the opinion of the investigator, could affect patient safety, preclude evaluation of response (e.g. because survival beyond 6 weeks is unlikely due to the underlying disease status)
10. Patient previously included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Overall survival 42 days | 42 days after the start of antifungal therapy
  Overall survival 42 days after the start of antifungal therapy in the MITT population

SECONDARY OUTCOMES:
Overall aspergillus attributable mortality | 12 weeks after the start of antifungal therapy
  Overall aspergillus attributable mortality 12 weeks after the start of antifungal therapy.
Overall survival 12 weeks | 12 weeks after the start of antifungal therapy
  Overall survival 12 weeks after the start of antifungal therapy in the MITT population
Overall survival 6 weeks (subgroup with positive serum galactomannan at baseline) | 6 weeks after the start of therapy
  Overall survival 6 weeks after the start of therapy in the subgroup of patients in the MITT population with a positive serum galactomannan test at baseline.
Overall survival 6 weeks (subgroup non-ICU patients who fulfill the EORTC/MSG probable or proven definition) | 6 weeks after the start of therapy
  Overall survival 6 weeks after the start of therapy in the subgroup of non-ICU patients who fulfill the EORTC/MSG probable or proven definition (MITT population).
Overall survival 6 weeks (subgroup of non-ICU patients with an underlying haematological disease (MITT population)) | 6 weeks after the start of therapy
  Overall survival 6 weeks after the start of therapy in the subgroup of non-ICU patients with an underlying haematological disease (MITT population)
Overall survival 6 weeks (subgroup of non-ICU patients without an underlying haematological disease (MITT population)) | 6 weeks after the start of therapy
  Overall survival 6 weeks after the start of therapy in the subgroup of non-ICU patients without an underlying haematological disease (MITT population)
Overall survival 6 weeks in patients that started with triazole monotherapy and in which triazole resistance is detected during follow-up (MITT population) | 6 weeks after the start of therapy
  Overall survival 6 weeks after the start of therapy in patients that started with triazole monotherapy and in which triazole resistance is detected during follow-up (MITT population)
Overall survival 6 weeks after the start of therapy in patients that started with triazole-anidulafungin combination therapy and in which triazole resistance is detected during follow-up (MITT population) | 6 weeks after the start of therapy
  Overall survival 6 weeks after the start of therapy in patients that started with triazole-anidulafungin combination therapy and in which triazole resistance is detected during follow-up (MITT population)
Kinetics of serum galactomannan levels | 6 weeks after the start of therapy
  In the subgroup of patients with a positive serum galactomannan; Kinetics of serum galactomannan levels with combination versus monotherapy
Mortality of patients in which resistance testing was unsuccessful | 12 weeks after the start of therapy
  Mortality of patients in which resistance testing was unsuccessful
Time to hospital discharge | 24 weeks after the start of therapy
  Time to hospital discharge (in the MITT subgroup of patients admitted to the hospital at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Belgium (2):
  - UZ Ghent, Ghent
  - UZ Leuven, Leuven
- Netherlands (2):
  - Erasmus Medical Center (EMC), Rotterdam, South Holland
  - Radboud Universitair Medisch Centrum, Nijmegen

REFERENCES:
- [Derived] Lamberink H, Huygens S, Aerts R, Lagrou K, van Leeuwen-Segarceanu E, Lodewyck T, Nieuwenhuizen L, Corsten MF, Moors I, Servais S, De Greef J, Hites M, Demandt A, Schauwvlieghe A, Maertens J, Rijnders B. Superiority Trials in Invasive Aspergillosis: A Harsh Reality Check With the IA-DUET (HOVON502) Trial. Clin Infect Dis. 2025 Feb 24;80(2):367-370. doi: 10.1093/cid/ciae501. PMID 39378343